CLINICAL TRIAL: NCT02335554
Title: Multimedia Internet-Based Program for Workers With Subthreshold Depression
Brief Title: Internet Program for Workers With Subthreshold Depression
Acronym: WorkDep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 81RR-2R
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Depression
Keywords: Subthreshold; Employees; Internet; Mobile; cognitive-behavioral
MeSH Terms: conditions — Depression | interventions — Workforce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MoodHacker (Experimental): Participants in the treatment condition were emailed a link to the MoodHacker mobile-web app and instructed to use the program for the next six weeks. Participants were asked to complete 2 follow-up assessments, 6 weeks and 10 weeks after baseline.
  Interventions: Behavioral: MoodHacker
- Alternative Care (Active Comparator): Alternative care participants were emailed and encouraged to browse links to vetted online information about depression. Participants were asked to complete 2 follow-up assessments, 6 weeks and 10 weeks after baseline and were given access to the MoodHacker program after the 10-week assessment
  Interventions: Behavioral: Alternative Care

INTERVENTIONS:
Behavioral: MoodHacker — Mobile-web app to educate users about depression and promote daily mood and positive activity monitoring.
  Other Names: Internet program for workers with subthreshold depression
  Arms: MoodHacker
Behavioral: Alternative Care — Online information about depression from government and other trusted sources to educate users about depression.
  Arms: Alternative Care

SUMMARY:
Depression is one of the most prevalent mental disorders to afflict adults. It seriously impacts role functioning and often takes a recurrent or chronic course. Because most adults who suffer from depression never receive treatment, there is a critical need to develop interventions that can be easily implemented and widely disseminated. Interventions that reduce the performance-impairing symptoms of subclinical depression and prevent the onset of major depression can improve employee well-being, while reducing healthcare costs and improving productivity. This project produced a mobile-web program to activate cognitive behavioral skills in workers with subthreshold depression, reduce depression symptoms, improve functioning in the workplace, and potentially reduce the risk for escalation to full-syndrome depression.

DETAILED DESCRIPTION:
The responsive mobile-web MoodHacker app was designed to: (a) educate users about depression; (b) educate users about the logistics and benefits of mood and activity monitoring; (c) promote daily mood and activity monitoring; (d) help users increase their positive activity engagement; (e) help users decrease negative thinking and increase positive thinking; and (f) promote daily practice of the skills taught.

Program content was adapted from the Coping with Depression group therapy course [18], enhanced with mindfulness-based [22] and other evidence-based positive psychology strategies [23-25]. Content for the application was refined based on input from experts in the field who had extensive experience working with adult employees at risk for depression. Additional program modifications were made based on data from individual interviews and iterative user testing with the population of interest during the formative and production phases of the project.

The MoodHacker user experience is structured around twelve learning objectives delivered through daily emails, in-app messaging, and in the "Articles & Videos" library. Daily emails (Figure 1) are sent to engage users in program content, provide sequenced guidance through the learning objectives in the articles and whiteboard-style videos, give tips for getting the most out of MoodHacker, and prompt the user to track their mood and activities daily. Users are encouraged to view the articles and videos as ordered, but viewing is not restricted, and users can view content according to their interest. The emails, articles and videos promote practice of the featured cognitive and behavioral skills outside the app experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* mild-to-moderate depressive symptoms as measured by the PHQ-9 (score of 10-19)
* not currently suicidal or meeting criteria for bipolar or schizo-affective disorder
* employed at least part-time
* English speaking
* access to a high-speed internet connection

Exclusion Criteria:

* younger than 18 years old
* severe depressive symptoms as measured by the PHQ-9 (score of 20+)
* currently suicidal or meeting criteria for bipolar or schizo-affective disorder
* employed less than part-time or unemployed
* not English speaking
* no access to a high-speed internet connection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Depression symptoms as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 10 week follow-up
  Depressive symptomatology was assessed at each assessment point using the self-reported Patient Health Questionnaire-9 scale to assess the nine DSM-IV major depression symptoms. The PHQ-9 is a self-report version of the Primary Care Evaluation of Mental Disorders (PRIME-MD) and has been shown to be a reliable and valid brief depression assessment tool.

SECONDARY OUTCOMES:
Activation of positive self-care and life-choice behaviors | 6-week posttest and 10-week follow-up
  How actively individuals are taking care of themselves, including making positive life choices, was expected to increase as a result of the intervention. Behavioral activation was measured using the Behavioral Activation for Depression Scale Short Form (BADS). This scale consists of 9 items.
Change in negative thinking | 6-week posttest and 10-week follow-up
  Change in negative thinking was assessed using the Automatic Thoughts Questionnaire - Revised scale Short Form (ATQ-R-SF). A 12-item adaptation of the ATQ-R instrument asked respondents to rate how many times over the past week they have had thoughts that are consistent with 12 negative self-statements.
Knowledge about depression | 6-week posttest and 10-week follow-up
  Treatment participants were assessed for an increase in knowledge about depression. The scale consisted of 14 multiple-choice items based on the 12 learning objectives addressed in the MoodHacker articles and videos.
Worker productivity as assessed by the Work Limitations Questionnaire | 6-week posttest and 10-week follow-up
  Worker productivity was assessed using the Work Limitations Questionnaire (WLQ). The WLQ Short Form consists of 10 items divided into four subscales measuring the degree to which a person was limited in their job's (1) time demands; (2) physical demands; (3) mental demands; and (4) output demands.
Worksite outcomes as assessed by the Workplace Outcomes Suite | 6-week posttest and 10-week follow-up
  Worksite outcomes were also assessed using the Workplace Outcomes Suite (WOS). The WOS is designed as an open-access instrument to facilitate empirical research on Employee Assistance Program (EAP) interventions. The suite contains five 5-item scales that assess: absenteeism, presenteeism, work engagement, life satisfaction, and workplace distress.
User satisfaction as assessed by the System Usability Scale | 6 week posttest
  Treatment participants completed the System Usability Scale, which is a quantitative measure of program ease of use. The scale includes 10 items. Users were asked to what degree they agreed or disagreed with program use and satisfaction statements on a 6-point scale (1=strongly disagree; 6=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Birney, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science

REFERENCES:
- [Derived] Birney AJ, Gunn R, Russell JK, Ary DV. MoodHacker Mobile Web App With Email for Adults to Self-Manage Mild-to-Moderate Depression: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2016 Jan 26;4(1):e8. doi: 10.2196/mhealth.4231. PMID 26813737